CLINICAL TRIAL: NCT06026241
Title: Practice Analysis of Care, Paraclinical Exams and Treatments Received by Geriatric Patients Both During the Last Week and the Last 24 Hours of Their Lives.
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1162023/CHUSTE
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: End-of-life Care
Keywords: End of life care; Geriatric; Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients over 75 who died in geriatrics: Patients over 75 years old who died in the geriatric short-stay departments of Saint-Etienne University Hospital
  Interventions: Other: Collecting data from the medical record

INTERVENTIONS:
Other: Collecting data from the medical record — Patient's socio-demographic data (age, gender, residence), comorbidities, cause of death, date and frequency of care measures/treatments/paraclinical exams received before their death.

SUMMARY:
End-of-life care is a core topic for geriatricians. One of the key aspects of end-of-life management is deciding when to discontinue active care measures (for example blood pressure monitoring, blood tests and X-rays) in favor of exclusive comfort care. In this retrospective observational study, the investigators looked at the care measures, treatments and paraclinical exams received by geriatric patients both one week and 24 hours before their death.

DETAILED DESCRIPTION:
This analysis provides information on the differences in geriatric physicians' practices regarding the anticipation of the end of life, by showing on average when active care measures were stopped before death. Secondly, the investigators looked at patient criteria that could explain a prolongation of active care and a delay in the implementation of exclusive comfort care.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 75 years old who died in a geriatric short-stay department at Saint-Etienne University Hospital.

Exclusion Criteria:

- Patients under 75 years old

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients over 75 years old who died in the geriatric short-stay departments of Saint-Etienne University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of care and treatments received during the last week of life, and during the last 24 hours of life | In the last week of life and 24 hours before death
  To measure the prevalence of care (hemodynamic, biological and radiological monitoring), and to evaluate the treatments received during the last week of life, and during the last 24 hours of life of patients hospitalized and who died in a geriatric short-stay ward.

SECONDARY OUTCOMES:
Patient criteria that may have explained the pursuit of care | In the last week of life and 24 hours before death
  Analysis of patient criteria (age, comorbidities, etc.) that may have explained the continuation of care, treatments and paraclinical exams up to the last 24 hours before death.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic LAFAIE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No